CLINICAL TRIAL: NCT02289274
Title: Partial Replicated Crossover Clinical Study to Compare Pharmacokinetic Characteristics of Eperisone and Aceclofenac With NVP-1203 Treatment to Those of Co-administration of Eperisone Hydrochloride Slow Release and Aceclofenac in Volunteers
Brief Title: Study to Compare Pharmacokinetic Characteristics of Eperisone and Aceclofenac With NVP-1203
Acronym: NVP-1203
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: internal decision
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1203-BE
Record Dates: First submitted 2014-11-09; First posted 2014-11-13 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — aceclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-1203 (Experimental): NVP-1203
  Interventions: Drug: NVP-1203
- Eperisone SR tab. + and Airtal tab. (Active Comparator): Eperisone HCl and aceclofenac
  Interventions: Drug: Eperisone SR tab. + and Airtal tab.

INTERVENTIONS:
Drug: NVP-1203 — NVP-1203(eperisone SR + aceclofenac)
  Other Names: Eperisone SR + aceclofenac
  Arms: NVP-1203
Drug: Eperisone SR tab. + and Airtal tab. — Eperisone SR and aceclofenac
  Other Names: Eperisone SR tab + airtal tab.
  Arms: Eperisone SR tab. + and Airtal tab.

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of NVP-1203 and coadministration of aceclofenac and eperisone HCl SR.

DETAILED DESCRIPTION:
aceclofenac and eperisone(low back pain)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age between 19 and 45
* BMI of >19kg/m2 and <28kg/m2 subject
* Informed of the investigational nature of this study and voluntarily agree to participate in this study

Exclusion Criteria:

* Use of any prescription medication within 14 days prior to Day 1
* Use of any medication within 7 days prior to Day 1

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve(AUC) last | 0-24hr

CONTACTS AND LOCATIONS:
Overall Officials: Bae K Seop, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Navipharm, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No